CLINICAL TRIAL: NCT01519843
Title: Post-stroke Procedural Learning: From Neural Substrates to Therapeutic Modulation by Non-invasive Brain Stimulation
Brief Title: Post Stroke Motor Learning
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Mont-Godinne (Other)
Responsible Party: Principal Investigator, Pr Yves Vandermeeren, MD, PhD, Professor, University Hospital of Mont-Godinne
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B039201212957
Record Dates: First submitted 2012-01-19; First posted 2012-01-27 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Stroke; Hemiparesis
Keywords: stroke
MeSH Terms: conditions — Stroke; Paresis | interventions — Transcranial Direct Current Stimulation; Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real (Active Comparator): Real tDCS
  Interventions: Device: transcranial direct current stimulation tDCS; Device: transcranial magnetic stimulation TMS
- sham (Placebo Comparator): Sham tDCS
  Interventions: Device: transcranial direct current stimulation tDCS; Device: transcranial magnetic stimulation TMS

INTERVENTIONS:
Device: transcranial direct current stimulation tDCS — tdcs (ELDITH, Neuroconn, Ilmenau, Germany)
Device: transcranial magnetic stimulation TMS — TMS (The Magstim Company Ltd, UK) Magstim 200² with a figure-of-eight coil was used to determine the hot spot eliciting consistent movements in the contralateral hand

SUMMARY:
Noninvasive brain stimulations (NIBS) will be used in chronic stroke patients to improve motor learning.

Functional magnetic resonance imaging will be used to evaluate the mechanisms underlying motor learning in healthy volunteers and in chronic stroke patients.

DETAILED DESCRIPTION:
transcranial direct current stimulation will be used for NIBS

ELIGIBILITY:
Inclusion Criteria:

* stroke with at least slight deficit

Exclusion Criteria:

* epilepsy
* contraindication to tDCS and/or to fMRI
* presence of metal in the head
* inability to understand / complete behavioral tasks
* chronic intake of alcohol or recreational drugs
* major health condition
* presence of pacemaker (for the fMRI part only)
* pregnancy

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Motor learning improvement with tDCS | Improvement on motor learning were recorded from baseline to 4 weeks after the intervention
  performance on a motor skill learning task and on different commonly used task (Purdue Pegboard, hand dynamometer, pinch dynamometer, 9-HPT ,...) were measured to explore the impact of tDCS on these parameters

SECONDARY OUTCOMES:
Neuroimaging | before motor learning, during motor learning and after (immediately, 30,60min) motor learning (with or without tDCS)
  Does cerebral mechanisms underlying motor learning differ from healthy subject to stroke patients?
Neurophysiological outcome measure | start of session 5min before motor learning, just at the end of the motor learning, after 30 min of motor learning, after 60 min of motor learning, Recall test at 1,2,3,4 weeks after the day of intervention (with or without tDCS)
  measure of brain excitability and connectivity with TMS (single and paired pulse)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, CHU Mont-Godinne, Yvoir, Namur, Belgium

REFERENCES:
- [Derived] Riga A, Gathy E, Ghinet M, De Laet C, Bihin B, Regnier M, Leeuwerck M, De Coene B, Dricot L, Herman B, Edwards MG, Vandermeeren Y. Evidence of Motor Skill Learning in Acute Stroke Patients Without Lesions to the Thalamus and Internal Capsule. Stroke. 2022 Jul;53(7):2361-2368. doi: 10.1161/STROKEAHA.121.035494. Epub 2022 Mar 21. PMID 35311345
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411